CLINICAL TRIAL: NCT05877911
Title: Effect of Sodium Thiosulfate on Nephrotoxicity of Cisplatin Intraperitoneal Heat-perfusion Chemotherapy: a Multi-center Prospective Randomized Controlled Trial.
Brief Title: Effect of Sodium Thiosulfate on Nephrotoxicity of Cisplatin Intraperitoneal Heat-perfusion Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Yunnan Cancer Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-549-02
Record Dates: First submitted 2023-04-03; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2022-11

CONDITIONS: Epithelial Ovarian Cancer; Acute Kidney Injury Due to Circulatory Failure
Keywords: Epithelial Ovarian Cancer; Acute Kidney Injury; Hyperthermic Intraperitoneal Chemotherapy; Sodium thiosulfate
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Acute Kidney Injury | interventions — sodium sulfate; Cisplatin

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to treatment group or control group by block randomisation in a 1:1 ratio.
  Treatment group: Receive HIPEC using sodium thiouracil and hydration Control group: Receive HIPEC only using hydration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIPEC with sodium thiosulfate and hydration (Experimental): Sodium sulfate 9 g/m^2 combined with 0.9% natrium chloride 150 ml were instilled in 20 min as the time when HIPEC with cisplatin was beginning. After that, sodium sulfate 12 g/m^2 combined with 0.9% natrium chloride 1000 ml was pumped for 6 h .
  hydration: On the day of surgery, the day of HIPEC, and 24 hours after HIPEC, daily intravenous rehydration should be performed using natrium chloride, glucose chloride or potassium chloride. The amount of fluid to be replenished should not be less than 3000 milliliters.
  Interventions: Drug: Sodium Sulfate; Other: Hydration; Drug: Cisplatin
- HIPEC with hydration only (Active Comparator): hydration:On the day of surgery, the day of HIPEC, and 24 hours after HIPEC, daily intravenous rehydration should be performed using natrium chloride, glucose chloride or potassium chloride. The amount of fluid to be replenished should not be less than 3000 milliliters.
  Interventions: Other: Hydration; Drug: Cisplatin

INTERVENTIONS:
Drug: Sodium Sulfate — Sodium thiosulfate has previously been reported to reduce the incidence of acute kidney injury after HIPEC with cisplatin, but this finding has not been confirmed in a high-level study.
  Arms: HIPEC with sodium thiosulfate and hydration
Other: Hydration — On the day of surgery, the day of HIPEC, and 24 hours after HIPEC, daily intravenous rehydration should be performed using natrium chloride, glucose chloride or potassium chloride. The amount of fluid to be replenished should not be less than 3000 milliliters.
Drug: Cisplatin — Infuse cisplatin (75mg/m^2) at 43℃ through the two drainage tubes placed in the upper abdomen, using the two drainage tubes placed in the lower abdomen as the effluent tubes, with an infusion time of 60-90 minutes and an infusion rate of 500-600 mL/min. The first HIPEC should be performed within 24-48 hours after cytoreductive surgery. The second HIPEC should be performed 24 hours after the completion of the first HIPEC. Intravenous sedatives such as dexmedetomidine or propofol at 2-6 ml/h should be administered during HIPEC treatment with continuous intravenous infusion by a pump，or intramuscular injection of 50 mg of pethidine.

SUMMARY:
Ovarian cancer is the most lethal malignancy of the female genital tract. Cytoreductive surgery combined with chemotherapy is the primary treatment for ovarian cancer, and radical tumor resection is an important means to improve the prognosis. However, even after complete tumor resection, 75% of patients with ovarian cancer still recur within 3 years after the initial treatment and eventually die from recurrence. In ovarian cancer, the lesions are located primarily in the peritoneal cavity. High-grade evidence demonstrates that the use of intraperitoneal hyperthermic chemotherapy (HIPEC) with cisplatin after cytoreductive surgery significantly improves the outcome in some patients with ovarian cancer. Currently, this is the only non-pharmacologic treatment that reduces both the risk of recurrence and death from ovarian cancer with a multi treatment. However, HIPEC with cisplatin can lead to acute kidney injury, and a serious complication that can seriously affect the short and long-term prognosis of patients. Sodium thiosulfate has previously been reported to reduce the incidence of acute kidney injury after HIPEC with cisplatin, but this finding has not been confirmed in a high-level study. Therefore, we propose a multi-center, prospective, open-label, randomized, controlled trial including 110 patients with ovarian cancer who received HIPEC with cisplatin, to evaluate whether sodium thiosulfate combined with hydration (55 patients in the trial group) can reduce the incidence of acute kidney injury after HIPEC with cisplatin compared with hydration alone (55 patients in the control group), and to provide high-level evidence for the rationale of using sodium thiosulfate for nephrotoxicity relief in cisplatin HIPEC.

ELIGIBILITY:
Inclusion Criteria:（The following conditions must be met at the same time）

* Patients treated with HIPEC with cisplatin.
* Estimated survival > 12 weeks
* Age from 18 to 70 years
* Bone marrow reserve was well functioning. Leukocytosis ≥ 3.0×10^9/L, neutrophilic granulocyte ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L, and hemoglobin ≥ 80 g/L.
* Organs work well. AST ≤ 2.5 × ULN, ALT ≤ 2.5 × upper limit of normal(ULN), total serum bilirubin ≤ 1.5 × ULN, and creatinine ≤ 1.5 × ULN
* ECOG score 0-1
* Patients voluntarily sign an informed consent form

Exclusion Criteria:（None of which was eligible）.

* Extensive abdominal adhesions
* HIPEC with Cisplatin for other medical conditions in the last 5 years.
* Receiving other drugs that cause kidney damage.
* Simultaneous use of amifotin for other diseases.
* Any situation of disease instability or potentially impact safety and adherence of patient.
* Chronic or acute nephropathy of any degree or other serious medical complications.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Calculate the incidence of acute kidney injury after HIPEC based on creatinine levels and 24-hour urine output according to KDIGO criteria. | Within one week after patients receive cisplatin-based HIPEC.
  To determine whether the use of sodium sulfate combined with hydration reduces the incidence of acute kidney injury (KDIGO criteria grade 1-3) effectively in the intention to treat population compared with hydration alone in patients receiving HIPEC with cisplatin (75mg/m^2,43 °C,90 minutes) according to creatinine levels and 24-hour urine.

SECONDARY OUTCOMES:
Calculate the incidence of chronic kidney injury after HIPEC based on creatinine levels according to KDIGO criteria. | Through study completion, an average of 2 year
  To determine whether the use of sodium sulfate combined with hydration reduces the incidence of chronic kidney injury effectively in the intention to treat population compared with hydration alone in patients receiving HIPEC with cisplatin (75mg/m^2,43 °C,90 minutes) according to creatinine levels.
Number of patients with sodium sulfate-related adverse events assessed by CTCAE v5.0. | 72 hours after sodium sulfate administration.
  To investigate adverse events associated with sodium sulfate. The Adverse events were evaluated and graded according to CTCAE5.0
Time from randomization to relapse or death（DFS）. | From date of randomisation to date of first recorded progression or death from any cause, whichever came first, assessed up to 5 years.
  Time from randomization to relapse or death. The diagnosis of disease recurrence includes CA125 more than two times the minimum value, as specified by the Gynecologic Cancer International Collaborative Group (GCIG), or according to the RECIST v1.1 criteria. Any one of the above two criteria is met first, then the tumor is recurrent.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong DK, Alvarez RD, Bakkum-Gamez JN, Barroilhet L, Behbakht K, Berchuck A, Chen LM, Cristea M, DeRosa M, Eisenhauer EL, Gershenson DM, Gray HJ, Grisham R, Hakam A, Jain A, Karam A, Konecny GE, Leath CA, Liu J, Mahdi H, Martin L, Matei D, McHale M, McLean K, Miller DS, O'Malley DM, Percac-Lima S, Ratner E, Remmenga SW, Vargas R, Werner TL, Zsiros E, Burns JL, Engh AM. Ovarian Cancer, Version 2.2020, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2021 Feb 2;19(2):191-226. doi: 10.6004/jnccn.2021.0007. PMID 33545690
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Kehoe S, Bhatla N. FIGO Cancer Report 2021. Int J Gynaecol Obstet. 2021 Oct;155 Suppl 1:5-6. doi: 10.1002/ijgo.13882. No abstract available. PMID 34669207
- [Background] Zivanovic O, Chi DS, Filippova O, Randall LM, Bristow RE, O'Cearbhaill RE. It's time to warm up to hyperthermic intraperitoneal chemotherapy for patients with ovarian cancer. Gynecol Oncol. 2018 Dec;151(3):555-561. doi: 10.1016/j.ygyno.2018.09.007. Epub 2018 Sep 22. PMID 30249527
- [Background] Lemoine L, Sugarbaker P, Van der Speeten K. Drugs, doses, and durations of intraperitoneal chemotherapy: standardising HIPEC and EPIC for colorectal, appendiceal, gastric, ovarian peritoneal surface malignancies and peritoneal mesothelioma. Int J Hyperthermia. 2017 Aug;33(5):582-592. doi: 10.1080/02656736.2017.1291999. PMID 28540826
- [Background] Lim MC, Chang SJ, Park B, Yoo HJ, Yoo CW, Nam BH, Park SY; HIPEC for Ovarian Cancer Collaborators. Survival After Hyperthermic Intraperitoneal Chemotherapy and Primary or Interval Cytoreductive Surgery in Ovarian Cancer: A Randomized Clinical Trial. JAMA Surg. 2022 May 1;157(5):374-383. doi: 10.1001/jamasurg.2022.0143. PMID 35262624
- [Background] Antonio CCP, Alida GG, Elena GG, Rocio GS, Jeronimo MG, Luis ARJ, Anibal ND, Francisco BV, Jesus GRA, Pablo RR, Jose GM. Cytoreductive Surgery With or Without HIPEC After Neoadjuvant Chemotherapy in Ovarian Cancer: A Phase 3 Clinical Trial. Ann Surg Oncol. 2022 Apr;29(4):2617-2625. doi: 10.1245/s10434-021-11087-7. Epub 2021 Nov 23. PMID 34812982
- [Background] Charo LM, Jou J, Binder P, Hohmann SF, Saenz C, McHale M, Eskander RN, Plaxe S. Current status of hyperthermic intraperitoneal chemotherapy (HIPEC) for ovarian cancer in the United States. Gynecol Oncol. 2020 Dec;159(3):681-686. doi: 10.1016/j.ygyno.2020.09.022. Epub 2020 Sep 22. PMID 32977989
- [Background] Furman MJ, Picotte RJ, Wante MJ, Rajeshkumar BR, Whalen GF, Lambert LA. Higher flow rates improve heating during hyperthermic intraperitoneal chemoperfusion. J Surg Oncol. 2014 Dec;110(8):970-5. doi: 10.1002/jso.23776. Epub 2014 Aug 29. PMID 25171494
- [Background] Liesenfeld LF, Wagner B, Hillebrecht HC, Brune M, Eckert C, Klose J, Schmidt T, Buchler MW, Schneider M. HIPEC-Induced Acute Kidney Injury: A Retrospective Clinical Study and Preclinical Model. Ann Surg Oncol. 2022 Jan;29(1):139-151. doi: 10.1245/s10434-021-10376-5. Epub 2021 Jul 14. PMID 34260006
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Hod T, Freedberg KJ, Motwani SS, Chen M, Frendl G, Leaf DE, Gupta S, Mothi SS, Richards WG, Bueno R, Waikar SS. Acute kidney injury after cytoreductive surgery and hyperthermic intraoperative cisplatin chemotherapy for malignant pleural mesothelioma. J Thorac Cardiovasc Surg. 2021 Apr;161(4):1510-1518. doi: 10.1016/j.jtcvs.2020.05.033. Epub 2020 May 29. PMID 32631662
- [Background] Chan CY, Li H, Wu MF, Liu CH, Lu HW, Lin ZQ, Li J. A Dose-Finding Trial for Hyperthermic Intraperitoneal Cisplatin in Gynecological Cancer Patients Receiving Hyperthermic Intraperitoneal Chemotherapy. Front Oncol. 2021 Mar 11;11:616264. doi: 10.3389/fonc.2021.616264. eCollection 2021. PMID 33777754
- [Background] Sin EI, Chia CS, Tan GHC, Soo KC, Teo MC. Acute kidney injury in ovarian cancer patients undergoing cytoreductive surgery and hyperthermic intra-peritoneal chemotherapy. Int J Hyperthermia. 2017 Sep;33(6):690-695. doi: 10.1080/02656736.2017.1293304. Epub 2017 Mar 5. PMID 28540777
- [Background] Cata JP, Zavala AM, Van Meter A, Williams UU, Soliz J, Hernandez M, Owusu-Agyemang P. Identification of risk factors associated with postoperative acute kidney injury after cytoreductive surgery with hyperthermic intraperitoneal chemotherapy: a retrospective study. Int J Hyperthermia. 2018 Aug;34(5):538-544. doi: 10.1080/02656736.2017.1368096. Epub 2017 Aug 29. PMID 28812384
- [Result] Colombo N, Sessa C, du Bois A, Ledermann J, McCluggage WG, McNeish I, Morice P, Pignata S, Ray-Coquard I, Vergote I, Baert T, Belaroussi I, Dashora A, Olbrecht S, Planchamp F, Querleu D; ESMO-ESGO Ovarian Cancer Consensus Conference Working Group. ESMO-ESGO consensus conference recommendations on ovarian cancer: pathology and molecular biology, early and advanced stages, borderline tumours and recurrent diseasedagger. Ann Oncol. 2019 May 1;30(5):672-705. doi: 10.1093/annonc/mdz062. PMID 31046081
- [Result] van Driel WJ, Koole SN, Sikorska K, Schagen van Leeuwen JH, Schreuder HWR, Hermans RHM, de Hingh IHJT, van der Velden J, Arts HJ, Massuger LFAG, Aalbers AGJ, Verwaal VJ, Kieffer JM, Van de Vijver KK, van Tinteren H, Aaronson NK, Sonke GS. Hyperthermic Intraperitoneal Chemotherapy in Ovarian Cancer. N Engl J Med. 2018 Jan 18;378(3):230-240. doi: 10.1056/NEJMoa1708618. PMID 29342393
- [Result] Kurreck A, Gronau F, Alberto Vilchez ME, Abels W, Enghard P, Brandl A, Francis R, Fohre B, Lojewski C, Pratschke J, Thuss-Patience P, Modest D, Rau B, Feldbrugge L. Sodium Thiosulfate Reduces Acute Kidney Injury in Patients Undergoing Cytoreductive Surgery Plus Hyperthermic Intraperitoneal Chemotherapy with Cisplatin: A Single-Center Observational Study. Ann Surg Oncol. 2022 Jan;29(1):152-162. doi: 10.1245/s10434-021-10508-x. Epub 2021 Aug 4. PMID 34350529
- [Result] Laplace N, Kepenekian V, Friggeri A, Vassal O, Ranchon F, Rioufol C, Gertych W, Villeneuve L, Glehen O, Bakrin N. Sodium thiosulfate protects from renal impairement following hyperthermic intraperitoneal chemotherapy (HIPEC) with Cisplatin. Int J Hyperthermia. 2020;37(1):897-902. doi: 10.1080/02656736.2020.1795277. PMID 32689832